CLINICAL TRIAL: NCT04868071
Title: Effects of Low-Speed and High-Speed Resistance Training Programs on Frailty Status, Physical Performance, Cognitive Function, and Blood Pressure in Prefrail and Frail Older Adults
Brief Title: Effects of Low-Speed and High-Speed Resistance Training Programs on Frailty Status
Acronym: RTF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Hélio José Coelho Júnior, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20021919.7.0000.5404
Record Dates: First submitted 2021-04-22; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Speed Resistance Training (Experimental): Participants performed exercises 8 times (sets) with 3-5 repetitions at 70%-75% of the maximal strength.
  Interventions: Behavioral: Physical Exercise
- Low-Speed Resistance Training (Experimental): Participants performed exercises 4 times (sets) with 8-10 repetitions at 70%-75% of the maximal strength.
  Interventions: Behavioral: Physical Exercise
- Control Group (No Intervention): No activities

INTERVENTIONS:
Behavioral: Physical Exercise — Exercise interventions were carried out over a total of 16 weeks in the mornings (08:00 am-12:00 am) under the supervision of at least two fitness instructors. Participants performed four exercises for lower limbs (Figure 9): 1st) squat on the chair, 2nd) seated unilateral hip flexion, 3rd) seated unilateral knee extension, and 4th) bilateral calf raise with 12-15 submaximal repetitions avoiding fatigue (i.e., inability to complete a repetition in a full range of motion). The number of sets was increased linearly during the first month, such that one set was performed in the 1st week, two sets in the 2nd week, 3 sets in the 3rd week, and 4 sets in the 4th week. Subsequently, participants performed the main exercise period. After a brief warm-up, participants performed the same exercises that were performed during the familiarization period using an adjustable weight vest and ankle weights (DOMYOS®, Shangai, China).
  Other Names: Resistance Training
  Arms: High-Speed Resistance Training; Low-Speed Resistance Training

SUMMARY:
The present study refers to a three-arm randomized controlled trial that investigated the effects of two types of RT on frailty status, physical performance, cognitive function, and blood pressure of prefrail and frail older adults.

ELIGIBILITY:
Inclusion Criteria:

* a) aged 60 years or over; b) were prefrail or frail according to Fried's criteria; c) performed the sit-to-stand test alone, with a mobility aid, or researcher's help; d) possessed sufficient physical and cognitive abilities to perform exercise sessions; and e) had a physician authorization to participate.

Exclusion Criteria:

* Exclusion criteria included having participated in a structured physical exercise training program in the past six months, prescription of hormone replacement therapy and/or psychotropic drugs, and any unstable cardiovascular event (e.g., myocardial infarction) or complication in the past 6 months.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Frailty Status | 16 weeks
  Frailty status will be assessed using the Fried Frailty Phenotype Scale published in 2001.
Physical Performance | 16 weeks
  Physical Performance will be assessed using the sit-to-stand test.
Cognitive Function | 16 weeks
  Cognition will be assessed using the Mini Mental State Examination
Blood Pressure | 16 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Cantinho do Idoso Senior Center, Poá, São Paulo
  - Mãe Maria Nursing Home, Poá, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coelho-Junior HJ, Uchida MC. Effects of Low-Speed and High-Speed Resistance Training Programs on Frailty Status, Physical Performance, Cognitive Function, and Blood Pressure in Prefrail and Frail Older Adults. Front Med (Lausanne). 2021 Jul 26;8:702436. doi: 10.3389/fmed.2021.702436. eCollection 2021. PMID 34381802